CLINICAL TRIAL: NCT03168152
Title: A Phase II Randomized Trial Comparing Stereotactic Body Radiation Therapy to Microwave Ablation for the Treatment of Localized Hepatocellular Carcinoma
Brief Title: Randomized Trial Comparing Stereotactic Body Radiation Therapy to Microwave Ablation for the Treatment of Localized Hepatocellular Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were accrued to the trial
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.001; HUM00124501 (Other: University of Michigan)
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWA (Experimental): MWA will typically be administered in one ablation session during which time up to 2 tumors are treated.
  Interventions: Radiation: Microwave Ablation (MWA)
- SBRT (Experimental): SBRT will be administered in five fractions of up to 10 Gy per fraction. SBRT will be administered 5-15 days per tumor.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Microwave Ablation (MWA) — MWA will typically be administered in one ablation session during which time up to 2 tumors are treated.
  Arms: MWA
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be administered in five fractions of up to 10 Gy per fraction. SBRT will be administered 5-15 days per tumor.
  Arms: SBRT

SUMMARY:
This is a randomized phase II study comparing microwave ablation (MWA) and stereotactic body radiation therapy (SBRT) for localized hepatocellular carcinoma (HCC).

This trial will be the first prospective comparison of these modalities for the treatment of HCC and will provide critical information regarding which local ablative modality is most appropriate for which patients. This study will also provide important information regarding quality of life and liver function changes following these two different treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma (HCC) are eligible for this trial. HCC is defined as having at least one of the following:

  1. HCC diagnosed either on biopsy or based on standard imaging criteria on contrast enhanced CT or MRI (arterial enhancement with washout and pseudocapsule); or
  2. A discrete hepatic tumor(s) as defined by the Barcelona criteria10 for cirrhotic patients, >1 cm with arterial hypervascularity and venous or delayed phase washout on CT or MRI
  3. Presentation at multidisciplinary liver tumor board to assess eligibility for either SBRT or MWA
* Patients must have 1-2 intrahepatic foci of HCC and may not be candidates for refuse hepatic resection. Patients who are on the organ wait list for (orthotopic liver transplantation) OLT will be considered for this trial as a "bridge" to transplant.
* Patients with 1 focus of HCC will be eligible if their tumor is 3.5 cm or less in greatest diameter. Patients with 2 foci of HCC will be eligible if each lesion is 3.5 cm in diameter or less and the combined diameter of both lesions is 5 cm or less.
* The foci of HCC must be in an anatomic location amendable to treatment by both MWA and SBRT.
* The patient must have an ECOG performance status of ≤ 2 (Eastern Cooperative Oncology Group Performance Status is an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death).
* Patients must have recovered from the acute effects of prior liver-directed therapy (e.g., RT, RFA, MWA or TACE) and a minimum of 4 weeks must have passed since the last procedure and protocol therapy.
* Patients must have:

  1. Platelets ≥ 50,000/mm3
  2. Child Pugh class A liver function or class B7 (Appendix II)
  3. INR (international normalized ratio (for anticoagulant monitoring)) < 1.5
* The patient must have a life expectancy of at least 12 weeks
* The patient must be at least 18 years old
* Patients must sign an IRB approved informed consent form for this purpose indicating that they are aware of the investigational aspects of the treatment and the potential risks. They also must be able to understand and the willing to sign a written informed consent.

Exclusion Criteria:

* Patients who have received prior abdominal radiation
* Patients with 3 or more foci of HCC
* Patients whose HCC involves the local vasculature, regional lymph nodes or distant metastatic sites
* Patients with Child Pugh liver function worse than B7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to local tumor progression | Patients will be followed up to 2 years
  The primary outcome of this trial is to prospectively determine local control rates in patients with HCC treated with MWA or SBRT. Freedom From Local Progression (FFLP) is defined as the time from randomization to local tumor progression. Tumors falling to group PD (progressive disease) would constitute local control failures. Progressive disease will be defined as at least a 20% increase in the LD (longest diameter) of target lesion, taking as reference the smallest LD recorded. Or at least a 20% increase in viable arterial enhancing disease, taking as reference the smallest LD of viable HCC since treatment started. Increases of less than 3 mm compared to the smallest LD recorded will be considered stable disease rather than PD.

SECONDARY OUTCOMES:
Incidence of gastrointestinal (GI) and hepatobiliary toxicity | Patients will be followed up to 2 years
  The number of patients experiencing grade 3 or higher GI or hepatobiliary toxicity by Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Incidence of liver function worsening | Patients will be followed up to 2 years
  The number of patients experiencing a 2 point or more increase in Child-Pugh score and an increase in albumin-bilirubin score of at least 0.5.
Change in FACT- Hep questionnaire score | Questionnaires will be administered pre-treatment, post-treatment, and at 1, 3 ,6, 9, 12, 15, 18, 21, and 24 months post-treatment
  The FACT-Hep questionnaire is used to measure health-related quality of life (HRQoL) in patients with hepatobiliary cancers. They are asked questions about their physical, social, emotional and functional well-being and asked to provide a score between 0 and 4 where 0 represents not at all and 4 represents very much.
Overall survival time | Patients will be followed up to 2 years
  Overall survival (OS) is defined as the time from randomization to death from any cause. Patients who are alive at last follow-up will be censored on that date.
Progression free survival time | Patients will be followed up to 2 years
  Progression Free Survival (PFS) is defined as the minimum time to death or any progression.
Metastasis free survival time | Patients will be followed up to 2 years
  Metastasis-free survival (MFS) is defined as the minimum time to development of metastases or death, whichever occurs first.
Incidence of intrahepatic failure | Patients will be followed up to 2 years
  Intrahepatic failure will include progression of the treated lesion(s) as well as development of other new liver lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Owen, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States